CLINICAL TRIAL: NCT05684484
Title: Clinical Study to Evaluate the Possible Efficacy and Safety of Roflumilast in Patients With Ulcerative Colitis.
Brief Title: Role of Roflumilast in Ulcerative Colitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, ahmed magdy youness, clinical pharmacist, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Roflumilast ulcerative colitis
Record Dates: First submitted 2022-12-26; First posted 2023-01-13 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Roflumilast; Tablets; Mesalamine

STUDY DESIGN:
Intervention Model Description: It will be conducted on 52 patient having with mild to moderate degree ulcerative colitis disease divided into two groups
  1. Placebo Group (n=26): Patients will receive conventional tratment only (amino salicylic acid) for 3 months.
  2. Group 2 (n=26): Patients will receive conventional treatment and Roflumilast (500 mcg ) orally once daily for 3 months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mesalamine group (Placebo Comparator): Placebo Group (n=26): Patients will receive mesalamine 500 mg once daily forulcerative colitis for 3 months.
  Interventions: Drug: amino salicylic acid
- Roflumilast group (Experimental): Patients will receive mesalamine and Roflumilast (500 mcg ) orally once daily for 3 months
  Interventions: Drug: Roflumilast 500 MCG Oral Tablet [DALIRESP]

INTERVENTIONS:
Drug: Roflumilast 500 MCG Oral Tablet [DALIRESP] — Roflumilast has been approved by U.S. Food and Drug Administration (FDA) for attenuating bronchial and dermatological disorders
  Other Names: phosphodiesterase type 4
  Arms: Roflumilast group
Drug: amino salicylic acid — conventional treatment
  Other Names: mesalamine
  Arms: mesalamine group

SUMMARY:
This study aims to investigate possible efficacy and safety of Roflumilast in adult patients with ulcerative colitis disease .

DETAILED DESCRIPTION:
* Study design and study population This study will be randomized, controlled, parallel study.
* It will be conducted on 52 patient having with mild to moderate degree ulcerative colitis disease divided into two groups

  1. Group 1 (n=26): Patients will receive conventional treatment only (corticosteroids +immune suppressive +amino salicylic acid) for 3 months.
  2. Group 2 (n=26): Patients will receive previous conventional treatment and Roflumilast (500 mcg ) orally once daily for 3 months
* Patient will be selected from Gastroenterology and Endoscopy Unit, Internal Medicine Department, Tanta University Hospital.
* A written informed consent will be obtained from all patients
* This study will be approved by the Research Ethics Committee of Tanta University.
* Any unexpected risks appeared during the course of research will be reported to the participants and ethical committee on time and documented through an adverse effects reporting form .
* Randomization will be carried out based on days of hospital admission

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to endoscopy units in Tanta University hospitals during the period of the study.

Patient with mild to moderate UC diagnosed as:

1. Clinical signs: Patients with moderate clinical disease have frequent loose, bloody stools (>4per day), mild anemia, and abdominal pain that is not severe. Patients have minimal signs of systemic toxicity, including a low-grade fever. Adequate nutrition is usually maintained, and weight loss.
2. Endoscopy : are necessary to establish the chronicity of inflammation and to exclude other causes of colitis.

Exclusion Criteria:

* Other inflammatory bowel disease (crohn's disease) .
* Patients <15 and >80 years
* Patients who didn't give consent to participate in the study
* Patients with contraindications of colonoscopy e.g. suspected colonic perforation, acute peritonitis, pregnancy, severe bleeding tendency, shock, uncooperative patient and if toxic mega colon is suspected were excluded
* History of allergic reaction to Roflumilast or any component of the formulation Like rash , hives ,itching and redness .
* Depression , thoughts of suicide , anxiety and emotional instability .
* Excessive weight loss .
* Moderate to severe hepatic impairment (child pugh class B or C) .
* Strong (CYP3A4) inducers : Barbiturates (phenobarbital) , Carbamazepine , Phenytoin , Rifampicin ( Risk , X interaction )
* Loxapine ( Risk , X interaction )

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
clinical improvement in ulcerative colitis severity | 3 months
  To demonstrate the efficacy of Roflumilast and clinical improvement in (Mayo disease activity index) for assessment of ulcerative colitis severity

SECONDARY OUTCOMES:
changes in serum levels of the measured biochemical parameters | 7 months
  demonstrate changes in serum levels of the measured biochemical parameters
  1. Tumor necrosis factor-alpha (TNF-α) as pro inflammatory marker (ELISA).
  2. Signal transducer and activator of transcription 3 (STAT3) as a potential marker for apoptosis ( ELISA)
  3. Caspase-3 as a potential marker for apoptosis (ELISA).

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of pharmacy Tanta university, Tanta, Egypt

REFERENCES:
- [Background] Feuerstein JD, Cheifetz AS. Ulcerative colitis: epidemiology, diagnosis, and management. Mayo Clin Proc. 2014 Nov;89(11):1553-63. doi: 10.1016/j.mayocp.2014.07.002. Epub 2014 Sep 8. PMID 25199861
- [Background] Thrash B, Patel M, Shah KR, Boland CR, Menter A. Cutaneous manifestations of gastrointestinal disease: part II. J Am Acad Dermatol. 2013 Feb;68(2):211.e1-33; quiz 244-6. doi: 10.1016/j.jaad.2012.10.036. PMID 23317981
- [Background] Neurath MF. Targeting immune cell circuits and trafficking in inflammatory bowel disease. Nat Immunol. 2019 Aug;20(8):970-979. doi: 10.1038/s41590-019-0415-0. Epub 2019 Jun 24. PMID 31235952
- [Background] de Souza HSP, Fiocchi C, Iliopoulos D. The IBD interactome: an integrated view of aetiology, pathogenesis and therapy. Nat Rev Gastroenterol Hepatol. 2017 Dec;14(12):739-749. doi: 10.1038/nrgastro.2017.110. Epub 2017 Aug 23. PMID 28831186
- [Background] Elbadry M, Nour MO, Hussien M, Ghoneem EA, Medhat MA, Shehab H, Galal S, Eltabbakh M, El-Raey F, Negm M, Afify S, Abdelhamed W, Sherief A, Abdelaziz A, Abo Elkasem M, Mahrous A, Kamal G, Maher M, Abdel-Hameed O, Elbasuny A, El-Zayyadi I, Bassiony A, Moussa A, Bedewy E, Elfert A, El Kassas M. Clinico-Epidemiological Characteristics of Patients With Inflammatory Bowel Disease in Egypt: A Nationwide Multicenter Study. Front Med (Lausanne). 2022 Apr 19;9:867293. doi: 10.3389/fmed.2022.867293. eCollection 2022. PMID 35514748
- [Background] Fujita Y, Khateb A, Li Y, Tinoco R, Zhang T, Bar-Yoseph H, Tam MA, Chowers Y, Sabo E, Gerassy-Vainberg S, Starosvetsky E, James B, Brown K, Shen-Orr SS, Bradley LM, Tessier PA, Ronai ZA. Regulation of S100A8 Stability by RNF5 in Intestinal Epithelial Cells Determines Intestinal Inflammation and Severity of Colitis. Cell Rep. 2018 Sep 18;24(12):3296-3311.e6. doi: 10.1016/j.celrep.2018.08.057. PMID 30232010
- [Background] Zundler S, Becker E, Schulze LL, Neurath MF. Immune cell trafficking and retention in inflammatory bowel disease: mechanistic insights and therapeutic advances. Gut. 2019 Sep;68(9):1688-1700. doi: 10.1136/gutjnl-2018-317977. Epub 2019 May 24. PMID 31127023
- [Background] Trivedi PJ, Adams DH. Chemokines and Chemokine Receptors as Therapeutic Targets in Inflammatory Bowel Disease; Pitfalls and Promise. J Crohns Colitis. 2018 Nov 28;12(12):1508. doi: 10.1093/ecco-jcc/jjy130. No abstract available. PMID 30272117
- [Background] Zhang X, Dong G, Li H, Chen W, Li J, Feng C, Gu Z, Zhu F, Zhang R, Li M, Tang W, Liu H, Xu Y. Structure-Aided Identification and Optimization of Tetrahydro-isoquinolines as Novel PDE4 Inhibitors Leading to Discovery of an Effective Antipsoriasis Agent. J Med Chem. 2019 Jun 13;62(11):5579-5593. doi: 10.1021/acs.jmedchem.9b00518. Epub 2019 May 31. PMID 31099559
- [Background] Raker VK, Becker C, Steinbrink K. The cAMP Pathway as Therapeutic Target in Autoimmune and Inflammatory Diseases. Front Immunol. 2016 Mar 31;7:123. doi: 10.3389/fimmu.2016.00123. eCollection 2016. PMID 27065076
- [Background] Li H, Li J, Zhang X, Feng C, Fan C, Yang X, Zhang R, Zhu F, Zhou Y, Xu Y, Liu H, Tang W. DC591017, a phosphodiesterase-4 (PDE4) inhibitor with robust anti-inflammation through regulating PKA-CREB signaling. Biochem Pharmacol. 2020 Jul;177:113958. doi: 10.1016/j.bcp.2020.113958. Epub 2020 Apr 3. PMID 32251674
- [Background] Li H, Fan C, Feng C, Wu Y, Lu H, He P, Yang X, Zhu F, Qi Q, Gao Y, Zuo J, Tang W. Inhibition of phosphodiesterase-4 attenuates murine ulcerative colitis through interference with mucosal immunity. Br J Pharmacol. 2019 Jul;176(13):2209-2226. doi: 10.1111/bph.14667. Epub 2019 May 17. PMID 30883697
- [Background] Zebda R, Paller AS. Phosphodiesterase 4 inhibitors. J Am Acad Dermatol. 2018 Mar;78(3 Suppl 1):S43-S52. doi: 10.1016/j.jaad.2017.11.056. Epub 2017 Dec 15. PMID 29248522
- [Background] Kokkonen K, Kass DA. Nanodomain Regulation of Cardiac Cyclic Nucleotide Signaling by Phosphodiesterases. Annu Rev Pharmacol Toxicol. 2017 Jan 6;57:455-479. doi: 10.1146/annurev-pharmtox-010716-104756. Epub 2016 Oct 12. PMID 27732797
- [Background] Faleiro L, Kobayashi R, Fearnhead H, Lazebnik Y. Multiple species of CPP32 and Mch2 are the major active caspases present in apoptotic cells. EMBO J. 1997 May 1;16(9):2271-81. doi: 10.1093/emboj/16.9.2271. PMID 9171342
- [Background] Kosutova P, Mikolka P, Kolomaznik M, Balentova S, Adamkov M, Calkovska A, Mokra D. Reduction of lung inflammation, oxidative stress and apoptosis by the PDE4 inhibitor roflumilast in experimental model of acute lung injury. Physiol Res. 2018 Dec 31;67(Suppl 4):S645-S654. doi: 10.33549/physiolres.934047. PMID 30607971